CLINICAL TRIAL: NCT02460016
Title: A Phase 1b, Open-label, Multicenter, Single Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of AK0529 in Infants Hospitalized With Respiratory Syncytial Virus Infection
Brief Title: A Study of AK0529 in Infants Hospitalized With RSV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We switched this study design to another study per IEC's recommendations.
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK0529-1002
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AK0529 (Experimental): AK0529 pellets
  Interventions: Drug: AK0529

INTERVENTIONS:
Drug: AK0529 — AK0529 pellets for oral administration
  Other Names: AK0529 pellets

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK) and anti-viral effect of single dose of AK0529 in infants hospitalized with respiratory syncytial virus (RSV).

DETAILED DESCRIPTION:
This is a open-label Phase 1b study to evaluate the safety, tolerability, pharmacodynamics and Pharmacokinetics of AK0529 in hospitalized RSV infected infants age from 1 to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race or ethnicity with an age adjusted for any prematurity of ≥1 month and ≤24 months.
* Diagnosis of RSV infection by virological.
* Subject must weigh >3 kg at screening.
* Must have provided written informed consent for the subject to participate.
* For patients aged <12 months, and occipitofrontal head circumference (OFHC) within the normal range for age and gender.

Exclusion Criteria:

* The subject has taken, is currently taking or requires any restricted medications.
* Subject is known to be HIV-positive (or the mother, if the potential subject is a child aged <6 months).
* Participation in an investigational drug or device study within 30 days prior to the date of screening.
* Requires vasopressors or inotropic support at the time of enrollment.
* Concurrent gastrointestinal conditions that could, in the opinion of the investigator, prejudice absorption of the Investigational Medicinal Product (e.g. protracted vomiting, malabsorption syndrome, a history of necrotising enterocolitis with consequent short gut syndrome).
* Bronchopulmonary dysplasia or chronic lung disease requiring assisted ventilation at the time of enrollment.
* Diminished ventilatory reserve at risk for hypercapnia (e.g. pulmonary hypoplasia, sequestration syndromes, cystadenomatoid malformation, a history of surgery for diaphragmatic hernia).
* Left to right shunt meriting corrective therapy.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2015-11-03 (Actual); Study Completion 2015-11-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Baseline through 7 days post administration

SECONDARY OUTCOMES:
Pharmacokinetics parameters, including maximum and minimum of drug concentration | Baseline through 3 days post administration
Pharmacokinetics parameters, including time to maximum concentration and half-time | Baseline through 3 days post administration
Pharmacokinetics parameters, including area under concentration-time curves (AUC) | Baseline through 3 days post administration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Toovey, MD PhD, Study Director — Shanghai Ark Biopharmaceutical Co., Ltd.
Locations (1):
- Women's & Children's Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No